CLINICAL TRIAL: NCT03689413
Title: Comparison of Sugammadex Dosages to Reverse the Effect of Rocuronium for Continuous Intraoperative Neuromonitoring in Thyroid Surgery
Brief Title: Adequate Dosage of Sugammadex on Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 30-2018-45
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Thyroid Surgery
Keywords: neuromonitoring; thyroid surgery
MeSH Terms: interventions — Sugammadex; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 mg/kg (Experimental): For '1 mg/kg' group, sugammadex of 1 mg/kg (ex. 60 mg for 60 kg patient) will be administered to the assigned patient for this group after tracheal intubation.
  We will use Sugammadex 200 MG in 2 ML Injection for this.
  Interventions: Drug: Sugammadex 200 MG in 2 ML Injection
- 2 mg/kg (Active Comparator): For '2 mg/kg' group, sugammadex of 2 mg/kg (ex. 120 mg for 60 kg patient) will be administered to the assigned patient for this group after tracheal intubation.
  We will use Sugammadex 200 MG in 2 ML Injection for this.
  Interventions: Drug: Sugammadex 200 MG in 2 ML Injection

INTERVENTIONS:
Drug: Sugammadex 200 MG in 2 ML Injection — 1 mg/kg or 2 mg/kg intravenous injection for each group (1 mg/kg group, 2 mg/kg group) after tracheal intubation
  Other Names: Bridion

SUMMARY:
This study was designed to compare two dosage of sugammadex after tracheal intubation for optimal condition of continuous intraoperative neuromonitoring in thyroid surgery to protect recurrent laryngeal nerve.

DETAILED DESCRIPTION:
Vocal cord paralysis is not a rare complication in thyroid surgery. Nerve monitoring technique has been developed, and many clinicians use the technique for saving the concerned nerves. Many studies showed that the effect of sugammadex on reverse of neuromuscular blocking after tracheal intubation. However, optimal dosage was not founded for sugammadex.

This randomized controlled trial is to compare 1 mg/kg and 2 mg/kg as dosage of sugammadex for optimal continuous intraoperative neuromonitoring in thyroid surgery to prevent vocal cord paralysis.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need to open thyroid surgery

Exclusion Criteria:

* Who doesn't agree to enroll
* Who has to receive other drug rather than rocuronium for muscle relaxant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Quality of signal of neuromonitoring | intraoperative
  During operation, surgeon evaluate the quality of signal of neuromonitoring on the basis of NIM III device.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- [Background] Empis de Vendin O, Schmartz D, Brunaud L, Fuchs-Buder T. Recurrent Laryngeal Nerve Monitoring and Rocuronium: A Selective Sugammadex Reversal Protocol. World J Surg. 2017 Sep;41(9):2298-2303. doi: 10.1007/s00268-017-4004-9. PMID 28349321
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Lu IC, Wu CW, Chang PY, Chen HY, Tseng KY, Randolph GW, Cheng KI, Chiang FY. Reversal of rocuronium-induced neuromuscular blockade by sugammadex allows for optimization of neural monitoring of the recurrent laryngeal nerve. Laryngoscope. 2016 Apr;126(4):1014-9. doi: 10.1002/lary.25577. Epub 2016 Jan 9. PMID 26748952